CLINICAL TRIAL: NCT02241473
Title: Changes in Body Composition, Metabolic and Mechanical Responses to Hypoxic Walking Training in Obese Patients
Brief Title: Hypoxic Training in Obese Patients
Acronym: HYPOBESE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lausanne (Other)
Collaborators: CHUV - Centre des Maladies Osseuses - Département de l'Appareil Locomoteur (DAL) (Unknown); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Davide MALATESTA, Dr (Ph.D., Senior Lecturer), University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136/14
Record Dates: First submitted 2014-09-10; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: gait; physical activity; energy cost; efficiency
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CH training group (Experimental): During 3 weeks (9 sessions; three sessions/wk), subject will performed 60 min walking at spontaneous walking speed in hypoxic (continuous hypoxic training, CHT; simulated altitude of 3000 m) condition in a single-blind fashion.
  Interventions: Other: Training
- CN training group (Active Comparator): During 3 weeks (9 sessions; three sessions/wk), subject will performed 60 min walking at spontaneous walking speed in normoxic (continuous normoxic training; CNT) condition in a single-blind fashion.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — During 3 weeks (9 sessions; three sessions/wk), subject will performed 60 min walking at spontaneous walking speed in normoxic (continuous normoxic training; CNT) or hypoxic (continuous hypoxic training, CHT; simulated altitude of 3000 m) condition in a single-blind fashion. Both CNT and CHT sessions will be performed in an hypoxic chamber (ATS Altitude, Sydney, Australia) built in our laboratory at an altitude of 380 m (Lausanne, Switzerland). In order to blind subjects to altitude, the system will also run for normoxic training groups with a normoxic airflow into the chamber.

SUMMARY:
By analyzing energetic and biomechanical basis of walking, and the subsequent changes induced by hypoxic vs normoxic training in obese individuals, it may optimize the use of walking in hypoxia to gain perspective for exercise prescription to set up training programs that aim to induce negative energy balance and to deal with weight management. However to the investigators knowledge, the analysis of changes in mechanics, energetics and efficiency of walking after continuous hypoxic training (CHT) has not been performed yet.

The aims of the present study were:

1. Comparing the changes in body composition between continuous hypoxic training (CHT) and similar training in normoxia; e.g. continuous normoxic training (CNT) in obese subjects.
2. Comparing the metabolic and energetics adaptations to CHT vs CNT.
3. Finally, comparing the associated body-loss induced gait modification since walking intensity at spontaneous walking speed (Ss) is lower in CHT than in CNT.

DETAILED DESCRIPTION:
Hypoxic training embraces different methods as "live high - train high" (LHTH) and "live high - train low" (LHTL); sleeping at altitude to gain the hematologic adaptations (increased erythrocyte volume) but training at sea level to maximize performance (maintenance of sea level training intensity and oxygen flux). The LHTL method can be accomplished via a number of methods and devices: natural/terrestrial altitude, nitrogen dilution, oxygen filtration and supplemental oxygen. Another method is the "live low - train high" (LLTH) method including intermittent hypoxic exposure at rest (IHE) or during intermittent hypoxic training sessions (IHT). Noteworthy, all supporting references were conducted with endurance elite athletes (i.e. cyclists, triathletes, cross-country skiers, runners, swimmers, kayakers, rowers) and there is an extensive literature relative both on LHTH and LHTL (Millet et al. 2010). Interestingly, very recently, the investigators research group proposed a new LLTH method (e.g. repeated sprints training in hypoxia; RSH) for team-sports players (Faiss et al. 2013). This lead to modify the nomenclature (Millet et al. 2013) and to divide LLTH method in four subsets; i.e. IHE, CHT (continuous >30 min low intensity training in hypoxia), IHT (interval-training in hypoxia) and RSH, based predominantly on different mechanisms; e.g. increased oxidative capacity (CHT), buffering capacity (IHT) or compensatory fiber-selective vasodilation (RSH). These new nomenclature and hypoxic methods open doors for investigating the use of different LLTH methods with other groups and for other purposes than the oxygen transport enhancement.

Several recent findings support the use of LLTH in obese subjects in terms of weight loss and/or cardiovascular and metabolic improvements (Kayser and Verges 2013). CHT [low intensity endurance exercise for 90 min at 60% of the heart rate at maximum aerobic capacity, 3 d week-1 for 8 weeks; fraction of inspired oxygen (FiO2) = 15%] in overweight subjects [body mass index (BMI) > 27] lead to larger (+1.1 kg) weight loss than similar training in normoxia. However, no difference was observed regarding BMI between the training modalities (Netzer et al. 2008). In a similar way, CHT (low intensity endurance exercise for 60 min at 65% of the heart rate at maximum aerobic capacity, 3 d week-1 for 4 weeks; FiO2 = 15%) induced similar increases in maximal oxygen consumption and endurance but larger improvements in respiratory quotient and lactate at the anaerobic threshold as well as in body composition than similar training in normoxia (Wiesner et al. 2010). Of interest is that the beneficial results were obtained despite lower training workload in hypoxia. This suggests that hypoxic training intensity can be lower in absolute value, at the spontaneous walking speed (Ss), also known as preferred or self-selected speed (e.g. the speed normally used during daily living activities). This appears to be an appropriate walking intensity for weight reduction programs aimed at inducing negative energy balance (Hills et al. 2006). A lower walking intensity is also likely more protective of the muscles/joints in obese patients with orthopaedic comorbidities. Finally, CHT was also shown (Haufe et al. 2008) to lead to larger change in body fat content, triglycerides, homeostasis assessment of insulin resistance (HOMA-Index), fasting insulin and area under the curve for insulin during an oral glucose tolerance test despite the lower absolute running intensity (1.4 and 1.7 W kg-1 in hypoxia and normoxia, respectively).

The net energy cost of level walking (NCw) represents the energy expenditure per distance unit only associated with walking movements. Previous studies reported higher absolute (J·m-1) and relative (i.e., normalized by body mass: J·kg-1·m-1) NCw in obese compared with normal body mass individuals (Browning et al. 2006; Peyrot et al. 2009), suggesting that the body mass is the main, but not the only, determinant of this lower economy of walking in obese subjects and that other factors may be involved in the higher NCw in these individuals(Browning et al. 2006; Peyrot et al. 2010; Peyrot et al. 2009). If body mass loss is an important method for the treatment of obesity and its associated co-morbidities and it may also be an important to investigate the effect of decreased body mass on gait pattern and mechanical external work (Wext) and their consequences on NCw in obese individuals. Walking is a fundamental movement pattern and the most common mode of physical activity. This form of locomotion may contribute significantly to weight management in overweight and obese subjects (Hill and Peters 1998; Jakicic et al. 2003; Pollock et al. 1971). Only one study showed that body mass reduction of 7% over 3 months resulted in gait kinematic changes (i.e., increases in walking speed, stride length and frequency, swing duration and decrease in cycle time, stance and double support time) in healthy adult obese women (BMI = 37 kg·m-2) (Plewa et al. 2007). However, these authors did not measure the NCw. More recently, Peyrot et al. (Peyrot et al. 2010) reported that, in healthy adolescent obese individuals, a 12-wk voluntary body mass reduction program (-6%) induced a reduction in NCw mainly associated with decreased body mass but also with changes in the biomechanical parameters of walking [i.e., a lesser lower limb muscle work required to rise the center of mass (CM) with Wext unchanged after intervention]. The authors hypothesized that the relation between the changes in absolute NCw and the changes in the biomechanical parameters might be explained by an increase in efficiency of muscle mechanical work with body mass loss as previously showed in cycling (Rosenbaum et al. 2003). Others studies (Messier et al. 2005; Messier et al. 2011), investigating only the effect of body mass loss (-3% and -10%, respectively) on biomechanical parameters of walking in non-healthy overweight and obese older adults with knee osteoarthritis, demonstrated that this body mass loss increased walking speed and reduced knee joint forces. Bariatric surgery may induce greater body mass loss (~30-40%) (Chaston et al. 2007) compared with exercise, diet or pharmaceutical interventions (~10%) (Franz et al. 2007) and may be considered as an interesting tool to maximize the effect of body mass loss on Wext and NCw in obese individuals and, thus, investigate the relationship between the gait pattern changes and the extra cost of walking in these subjects. Similarly, it would be of interest to investigate how the metabolic changes and body mass loss induced by CHT, potentially associated with an increased metabolic efficiency, would affect gait pattern and the extra cost of walking in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free of clinically significant orthopaedic, neurological, cardiovascular or respiratory conditions.
* BMI > 30 kg/m^2.
* Age > 18 yr.

Exclusion Criteria:

* Age > 40 yr.
* BMI < 35 kg/m^2.
* Diabetes.
* Neurological disorders, orthopaedic injury, history of falls and medications that provoke dizziness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Body composition and mass | Change from baseline at 5 weeks (e.g., baseline and 5th week after inclusion)
  All subjects will undergo dual-energy X-ray absorptiometry (DEXA) and bio-impedance for measurements of body composition.
Net energy cost of walking | Change from baseline at 5 weeks (e.g., baseline and 5th week after inclusion)
  The subjects will be then asked to complete five 6 min level walking trials on the instrumented treadmill at five equally spaced speeds (0.55, 0.83, 1.11, 1.38 and 1.66 m/s), in randomized order. They will be allowed to establish their own preferred stride rate combination for each condition and will be given 5 min of rest between walking trials. During the walking trials, oxygen uptake (V˙O 2), carbon dioxide (CO2) output (V˙C O2) and ventilation (V˙ E) will be measured breath-by-breath (OxyconPro, Jaeger, Germany) and the volume and gases calibrations will be checked before each trial. Oxygen uptake values from the last 2 min will be averaged and normalized to body mass (V˙O 2, mlO2∙kg-1∙min-1). This value minus resting V'O2 was then divided by walking speed to obtain the net energy cost of walking (mlO2∙kg-1∙m-1).
Mechanical external and internal work | Change from baseline at 5 weeks (e.g., baseline and 5th week after inclusion)
  During steady metabolic state (i.e., the last 2 min of walking for each speed), the mechanical external (Wext) and internal (Wint) work changes of 20 consecutive walking steps will be determined with an instrumented treadmill (H-P-COSMOS Treadmill MCU2 EPROM 2.31), consisting of a treadmill mounted on four 3-D force sensors, following the methods described in detail by Cavagna (Cavagna 1975) and Willems et al. (1995).
Efficiency | Change from baseline at 5 weeks (e.g., baseline and 5th week after inclusion)
  Total mechanical work and efficiency. The total mass-specific muscular work per distance travelled (Wtot) will be calculated as the sum of Wext and Wint. The mechanical efficiency will be computed as the ratio between Wtot and net energy cost of walking.

SECONDARY OUTCOMES:
Blood samples (this measure is a composite) | Change from baseline at 5 weeks (e.g., baseline and 5th week after inclusion)
  The blood samples were drawn at rest before (session 1) and after (session 12) the training program during fasting to determine total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL) and triglycerides (TG), leptin, total adiponectin, resistin, retinol-binding protein 4 (RBP4), plasma glucose and insulin concentrations (this measure is a composite).

CONTACTS AND LOCATIONS:
Overall Officials: Davide Malatesta, Dr, Principal Investigator — Institute of Sport Sciences of the University of Lausanne
Locations (1):
- Institute of Sport Sciences of the University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Browning RC, Baker EA, Herron JA, Kram R. Effects of obesity and sex on the energetic cost and preferred speed of walking. J Appl Physiol (1985). 2006 Feb;100(2):390-8. doi: 10.1152/japplphysiol.00767.2005. Epub 2005 Oct 6. PMID 16210434
- [Background] Faiss R, Leger B, Vesin JM, Fournier PE, Eggel Y, Deriaz O, Millet GP. Significant molecular and systemic adaptations after repeated sprint training in hypoxia. PLoS One. 2013;8(2):e56522. doi: 10.1371/journal.pone.0056522. Epub 2013 Feb 20. PMID 23437154
- [Background] Haufe S, Wiesner S, Engeli S, Luft FC, Jordan J. Influences of normobaric hypoxia training on metabolic risk markers in human subjects. Med Sci Sports Exerc. 2008 Nov;40(11):1939-44. doi: 10.1249/MSS.0b013e31817f1988. PMID 18845972
- [Background] Hill JO, Peters JC. Environmental contributions to the obesity epidemic. Science. 1998 May 29;280(5368):1371-4. doi: 10.1126/science.280.5368.1371. PMID 9603719
- [Background] Kayser B, Verges S. Hypoxia, energy balance and obesity: from pathophysiological mechanisms to new treatment strategies. Obes Rev. 2013 Jul;14(7):579-92. doi: 10.1111/obr.12034. Epub 2013 Mar 28. PMID 23551535
- [Background] Messier SP, Gutekunst DJ, Davis C, DeVita P. Weight loss reduces knee-joint loads in overweight and obese older adults with knee osteoarthritis. Arthritis Rheum. 2005 Jul;52(7):2026-32. doi: 10.1002/art.21139. PMID 15986358
- [Background] Messier SP, Legault C, Loeser RF, Van Arsdale SJ, Davis C, Ettinger WH, DeVita P. Does high weight loss in older adults with knee osteoarthritis affect bone-on-bone joint loads and muscle forces during walking? Osteoarthritis Cartilage. 2011 Mar;19(3):272-80. doi: 10.1016/j.joca.2010.11.010. Epub 2010 Dec 4. PMID 21134477
- [Background] Millet GP, Faiss R, Brocherie F, Girard O. Hypoxic training and team sports: a challenge to traditional methods? Br J Sports Med. 2013 Dec;47 Suppl 1(Suppl 1):i6-7. doi: 10.1136/bjsports-2013-092793. No abstract available. PMID 24282210
- [Background] Millet GP, Roels B, Schmitt L, Woorons X, Richalet JP. Combining hypoxic methods for peak performance. Sports Med. 2010 Jan 1;40(1):1-25. doi: 10.2165/11317920-000000000-00000. PMID 20020784
- [Background] Netzer NC, Chytra R, Kupper T. Low intense physical exercise in normobaric hypoxia leads to more weight loss in obese people than low intense physical exercise in normobaric sham hypoxia. Sleep Breath. 2008 May;12(2):129-34. doi: 10.1007/s11325-007-0149-3. PMID 18057976
- [Background] Peyrot N, Morin JB, Thivel D, Isacco L, Taillardat M, Belli A, Duche P. Mechanical work and metabolic cost of walking after weight loss in obese adolescents. Med Sci Sports Exerc. 2010 Oct;42(10):1914-22. doi: 10.1249/MSS.0b013e3181da8d1e. PMID 20216466
- [Background] Peyrot N, Thivel D, Isacco L, Morin JB, Duche P, Belli A. Do mechanical gait parameters explain the higher metabolic cost of walking in obese adolescents? J Appl Physiol (1985). 2009 Jun;106(6):1763-70. doi: 10.1152/japplphysiol.91240.2008. Epub 2009 Feb 26. PMID 19246657
- [Background] Plewa M, Cieślińska-Świder J, and Bacik B. Effects of the Weight loss Treatment on Selected Kinematic Gait Parameters in Obese Women. Journal of Human Kinetics 18: 3-14, 2007.
- [Background] Pollock ML, Miller HS Jr, Janeway R, Linnerud AC, Robertson B, Valentino R. Effects of walking on body composition and cardiovascular function of middle-aged man. J Appl Physiol. 1971 Jan;30(1):126-30. doi: 10.1152/jappl.1971.30.1.126. No abstract available. PMID 5538779
- [Background] Rosenbaum M, Vandenborne K, Goldsmith R, Simoneau JA, Heymsfield S, Joanisse DR, Hirsch J, Murphy E, Matthews D, Segal KR, Leibel RL. Effects of experimental weight perturbation on skeletal muscle work efficiency in human subjects. Am J Physiol Regul Integr Comp Physiol. 2003 Jul;285(1):R183-92. doi: 10.1152/ajpregu.00474.2002. Epub 2003 Feb 27. PMID 12609816
- [Background] Wiesner S, Haufe S, Engeli S, Mutschler H, Haas U, Luft FC, Jordan J. Influences of normobaric hypoxia training on physical fitness and metabolic risk markers in overweight to obese subjects. Obesity (Silver Spring). 2010 Jan;18(1):116-20. doi: 10.1038/oby.2009.193. Epub 2009 Jun 18. PMID 19543214
- [Derived] Fernandez Menendez A, Saudan G, Sperisen L, Hans D, Saubade M, Millet GP, Malatesta D. Effects of Short-Term Normobaric Hypoxic Walking Training on Energetics and Mechanics of Gait in Adults with Obesity. Obesity (Silver Spring). 2018 May;26(5):819-827. doi: 10.1002/oby.22131. Epub 2018 Mar 25. PMID 29575698